CLINICAL TRIAL: NCT03078647
Title: Clinical Study to Evaluate the Safety and Efficacy Performance of the Profound System Using the Dermal and Sub-dermal (SubQ) Cartridges for the Treatment of Cellulite
Brief Title: Profound Dermal and SubQ Cartridges for the Treatment of Cellulite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF21711
Record Dates: First submitted 2017-02-22; First posted 2017-03-13 (Actual); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Profound treatment to small areas (Experimental): Single Profound treatment with the Dermal and/or SubQ cartridges to bra bulge, above the knees or upper arms
  Interventions: Device: Profound

INTERVENTIONS:
Device: Profound — The main intent of the Profound Dermal and Subdermal cartridges for cellulite treatment is to utilize a minimally-invasive approach to directly deliver radiofrequency (RF) energy into tissue through pairs of micro-electrode needles and use temperature sensors within the needles to reliably create fractional thermal injuries within the skin.

SUMMARY:
Clinical Study to Evaluate the Performance of the Profound System for the Treatment of Cellulite.

DETAILED DESCRIPTION:
Up to 60 healthy female volunteers, seeking cellulite treatment, 18 to 60 years of age from up to 3 investigational sites.

Prospective, open-label, baseline-controlled, two arms, randomized, clinical study to evaluate the Profound device using the Dermal and SubQ Cartridges for minimally-invasive treatment of the upper thighs and buttocks cellulite appearance.

The treatment areas of the study subjects will be divided into two arms:

1. Arm 1 - the upper thigh/buttock on the left or right side of the body will undergo a single Profound treatment utilizing the Dermal and SubQ Cartridges
2. Arm 2 - the contralateral upper thigh/buttock side of the body will undergo a single Profound treatment utilizing the SubQ Cartridge only.

Methodology described in protocol to evaluate efficacy of treatments will be carried out at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Female subjects, ≥ 18 and ≤ 60 years of age at the time of enrollment
3. Fitzpatrick Skin Type I to VI.
4. Subjects seeking treatment of cellulite in the upper thighs and buttocks areas.
5. Subject cellulite stage II or III as graded using Nurnberger-Muller scale classification (Appendix III).
6. Not pregnant, lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. Negative urine pregnancy test as tested prior to each treatment and at the last visit for women of child bearing potential (e.g. not menopause).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to receive the proposed Profound treatment.
10. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
11. Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations.

Exclusion Criteria:

1. Subject cellulite stage 0 or I as graded using Nurnberger-Muller scale classification (Appendix III).
2. Subject had surgery or any other procedure for cellulite in the last 6 months.
3. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
4. Known allergy to lidocaine or epinephrine or antibiotics.
5. Active malignancy or history of malignancy in the past 5 years.
6. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
7. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders (i.e. any disease state that in the opinion of the Physician would interfere with the anesthesia, treatment, or healing process).
8. Having a known anti-coagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion).
9. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
10. Suffering from hormonal imbalance, whether related to thyroid, pituitary, or androgen.
11. History of significant lymphatic drainage problems.
12. History of cancer which required lymph node biopsy or dissection.
13. Suffering from significant skin conditions in treatment areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
14. History of keloid scarring, abnormal wound healing and / or prone to bruising.
15. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
16. Use of isotretinoin (Accutane) within 6 months of treatment or during the study.
17. Subject on systemic corticosteroid therapy 6 months prior to and throughout the course of the study.
18. Dysplastic nevi in the area to be treated.
19. Participation in a study of another device or drug within 3 month prior to enrollment or during this study.
20. Subject has palpable lymphadenopathy at any visit. Standard palpation techniques will be used.
21. Subjects with history of severe edema.
22. As per the Investigator's discretion, any physical or mental condition that might make it unsafe for subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Girish Munavalli, MD, Principal Investigator — Laser & Vein Specialists of the Carolinas
Locations (2):
- United States (2):
  - Macrene Alexiades, New York, New York
  - Girish Munavalli, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawlings AV. Cellulite and its treatment. Int J Cosmet Sci. 2006 Jun;28(3):175-90. doi: 10.1111/j.1467-2494.2006.00318.x. PMID 18489274
- [Background] Rossi AB, Vergnanini AL. Cellulite: a review. J Eur Acad Dermatol Venereol. 2000 Jul;14(4):251-62. doi: 10.1046/j.1468-3083.2000.00016.x. PMID 11204512
- [Background] Alexiades M, Berube D. Randomized, blinded, 3-arm clinical trial assessing optimal temperature and duration for treatment with minimally invasive fractional radiofrequency. Dermatol Surg. 2015 May;41(5):623-32. doi: 10.1097/DSS.0000000000000347. PMID 25915628
- [Background] Alexiades M, Munavalli G, Goldberg D, Berube D. Prospective Multicenter Clinical Trial of a Temperature-Controlled Subcutaneous Microneedle Fractional Bipolar Radiofrequency System for the Treatment of Cellulite. Dermatol Surg. 2018 Oct;44(10):1262-1271. doi: 10.1097/DSS.0000000000001593. PMID 30222637
- [Derived] Alexiades M, Munavalli GS. Single Treatment Protocol With Microneedle Fractional Radiofrequency for Treatment of Body Skin Laxity and Fat Deposits. Lasers Surg Med. 2021 Oct;53(8):1026-1031. doi: 10.1002/lsm.23397. Epub 2021 Mar 25. PMID 33764552

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated on the Suprapatellar: Subjects treated with the Profound Dermal, SubQ or both cartridges above the knees areas (on both left and right sides)
- Treated on the Upper Arms: Subjects treated with the Profound Dermal, SubQ or both cartridges on the upper arms (on both left and right sides)
- Treated on the Braline: Subjects treated with the Profound Dermal, SubQ or both cartridges on the braline areas (on both left and right sides)
Period: Overall Study
Arm/Group | Treated on the Suprapatellar | Treated on the Upper Arms | Treated on the Braline
Started | 17 | 11 | 3
Completed | 17 | 10 | 3
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects treated with Profound SubQ, Dermal or both cartridges. Each subject was treated in two contralateral areas. If each area was treated differently (e.g. different cartridge or parameters used) it was assessed separately.
Units Other Than Participants: Number Areas
Groups:
- Treated on the Suprapatellar: Subjects treated with the Profound Dermal, SubQ or both cartridges above the knees areas (on both the left and the right side)
- Treated on the Upper Arms: Subjects treated with the Profound Dermal, SubQ or both cartridges on the upper arms (on both the left and the right side)
- Treated on the Braline: Subjects treated with the Profound Dermal, SubQ or both cartridges on the braline areas (on both the left and the right side)
- Total: Total of all reporting groups
Arm/Group | Treated on the Suprapatellar | Treated on the Upper Arms | Treated on the Braline | Total
Number analyzed (Participants) | 17 | 11 | 3 | 31
Number analyzed (Number Areas) | 34 | 22 | 6 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 3 | 31
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (8.8) | 53.8 (6.8) | 46.7 (14.6) | 50.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 3 | 31
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 11 | 3 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 17 | 11 | 3 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 11 | 3 | 31

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Global Aesthetic Appearance of Cellulite in Treated Areas, as Assessed by Study Investigator Evaluations
Description: Evaluate the improvement in global aesthetic appearance of cellulite in treated areas following a single dermal and/or subcutaneous treatment with Profound, as assessed by study investigators at 1,3 and 6 months post treatment visit. Investigators used the following scale: 0=No Change; 1= 1-24% improvement; 2=25-49% improvement; 3=50-74% improvement; 4=75-100% improvement.
  The analysis calculates the improvement over 25% (grades 2-4)
Time Frame: 1,3 and 6 months post-treatment
Population: Suprapatellar areas- 17 subjects, 8 subjects (16 areas) had one assessment for both sides treated with the same parameters.
  Upper Arms- 10 Subjects had one assessment for both sides treated with same parameters (1 subject dropped after 1 wk FU).
  Braline areas- 3 subjects, one subject had one assessment for both sides treated with same parameters
Measure: Count of Units; unit: Investigator Assessments
Units Other Than Participants: Investigator Assessments
Arm/Group | Treated on the Suprapatellar | Treated on the Upper Arms | Treated on the Braline
Number analyzed (Participants) | 17 | 10 | 3
Number analyzed (Investigator Assessments) | 26 | 10 | 5
Investigator Assessments
  Over 25% Improvement at 1 month FU | 11 | 7 | 4
  Over 25% Improvement at 3 month FU | 16 | 10 | 5
  Over 25% Improvement at 6 month FU | 15 | 9 | 4

2. Secondary Outcome: Improvement in Skin Tightening/Laxity in Treated Areas, as Assessed by Study Investigator Evaluations
Description: Evaluate the improvement in skin tightening in treated areas following a single dermal and/or subcutaneous treatment with Profound, as assessed by study investigators at 1 and 6 months post treatment visit. Investigators used the following scale: (0) No tightening/firmness; (1) Slightly visible tightening/firmness; (2) Visible tightening/firmness; (3) Very visible tightening/firmness.
  The analysis calculates the skin tightening improvement graded: (2) Visible tightening/firmness and (3) Very visible tightening/firmness
Time Frame: 1, 3 and 6 months post treatment visit.
Population: as for outcome 1
Measure: Count of Units; unit: Investigator Assessments
Units Other Than Participants: Investigator Assessments
Arm/Group | Treated on the Suprapatellar | Treated on the Upper Arms | Treated on the Braline
Number analyzed (Participants) | 17 | 10 | 3
Number analyzed (Investigator Assessments) | 26 | 10 | 5
Investigator Assessments
  Visible + very visible tightening at 1-month FU | 9 | 3 | 4
  Visible + very visible tightening at 3-month FU | 14 | 8 | 4
  Visible + very visible tightening at 6-month FU | 15 | 8 | 4

3. Secondary Outcome: Investigator Satisfaction - by Questionnaire
Description: Evaluate Investigator satisfaction at 1, 3, and 6 months post-treatment visit, using a satisfaction scale [(-2) Very dissatisfied, (-1) Dissatisfied, (0) No opinion, (1) Satisfied, (2) Very satisfied].
  The analysis quantify investigator satisfaction (grades 1-2)
Time Frame: 1, 3, and 6 months post-treatment visit
Population: as for outcome 1
Measure: Count of Units; unit: Investigator Assessments
Units Other Than Participants: Investigator Assessments
Arm/Group | Treated on the Suprapatellar | Treated on the Upper Arms | Treated on the Braline
Number analyzed (Participants) | 17 | 10 | 3
Number analyzed (Investigator Assessments) | 26 | 10 | 5
Investigator Assessments
  Investigator Satisfaction Grades 1-2 at 1mo FU | 13 | 8 | 4
  Investigator Satisfaction Grades 1-2 at 3mo FU | 21 | 10 | 4
  Investigator Satisfaction Grades 1-2 at 6mo FU | 17 | 9 | 4

4. Secondary Outcome: Subject Satisfaction and Improvement - by Questionnaire
Description: Evaluate subject satisfaction at 1, 3, and 6 months post-treatment visit, using a satisfaction and improvement scale [(-2) Very dissatisfied, (-1) Dissatisfied, (0) No opinion, (1) Satisfied, (2) Very satisfied].
  The analysis quantify subject satisfaction (grades 1-2)
Time Frame: 1, 3, and 6 months post-treatment visit
Population: as for outcome 1
Measure: Count of Units; unit: Subject Assessments
Units Other Than Participants: Subject Assessments
Arm/Group | Treated on the Suprapatellar | Treated on the Upper Arms | Treated on the Braline
Number analyzed (Participants) | 17 | 10 | 3
Number analyzed (Subject Assessments) | 26 | 10 | 5
Subject Assessments
  Subject Satisfaction Grades 1-2 at 1mo FU | 13 | 8 | 2
  Subject Satisfaction Grades 1-2 at 3mo FU | 20 | 10 | 2
  Subject Satisfaction Grades 1-2 at 6mo FU | 17 | 10 | 4

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected is from treatment visit until 6 month post treatment
Description: The number and severity of adverse events following a single dermal and subcutaneous treatment, with Profound for the Suprapatellar, upper arms or braline, were evaluated at 1-week post treatment, 1 month, 3 and 6 months following the treatment.
Arm/Group | Treated on the Suprapatellar | Treated on the Upper Arms | Treated on the Braline
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/11 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 1/17 | 0/11 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated on the Suprapatellar (N=17) | Treated on the Upper Arms (N=11) | Treated on the Braline (N=3)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild bruising reported on 1 week FU visit, located at the right knee. Recovered after 2 days without intervention.
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild itching reported at the 1 week FU, located at the right and left knees. Recovered after 2 days without intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT03078647/Prot_SAP_000.pdf